CLINICAL TRIAL: NCT06113094
Title: Cryoablation for Advanced and Refractory Desmoid Tumors
Acronym: CARDT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7884
Record Dates: First submitted 2022-11-14; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2022-11

CONDITIONS: Desmoid Tumors
Keywords: Desmoid tumors; Fibromatosis; Invasive tumors; Radiotherapy; Cryoablation
MeSH Terms: conditions — Desmoid Tumors; Fibroma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Desmoid tumors, also called aggressive fibromatosis, are rare, locally invasive tumors with no potential for metastasis. The incidence is approximately 2 to 4 per million per year in the general population. The "watch and wait" policy is the standard of care for newly diagnosed patients in Europe. Patients who progress have first-line medical treatment, surgery is no longer the treatment because there is a high rate of recurrence (> 60%) and radiotherapy is not very suitable because the patients are often young and the tumors are large. Cryoablation seems to be an effective therapeutic option that should be evaluated.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Having undergone cryoablation for an advanced desmoid tumor refractory to medical treatment
* Having not expressed their opposition, after being informed, to the reuse of their data for the purposes of this research.

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Patient already included in another ongoing study
* Subject under guardianship or curatorship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) having undergone cryoablation for an advanced desmoid tumor refractory to medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival assessed using RECIST(Response evaluation criteria in solid tumors) criteria | at 6 months after cryoablation

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Imagerie Interventionnelle - CHU de Strasbourg - France, Strasbourg, France